CLINICAL TRIAL: NCT04206462
Title: Investigation of Oxidative Markers and Antioxidant Defense in Female Patients With Osteoarthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Rodica Ana Ungur, Principal investigator, Iuliu Hatieganu University of Medicine and Pharmacy
Other Study IDs: UniversitateaIH
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Osteoarthritis: Questionnaire of eating habits, markers of oxidative stress
  Interventions: Other: Questionnaire of eating habits

INTERVENTIONS:
Other: Questionnaire of eating habits — frequency and type of aliments

SUMMARY:
Osteoarthritis has a multifactorial etiology: aging, genetic, sex, weight, alimentation, injuries, infections etc. The objective of the study is to investigate the eating behaviour of the patients included in the study by using a semiquantitative questionnaire (frequency and quantity) by estimating the foods that are known to be protective for osteoarthritis (vegetables, fruits, cereals) as the ones that are considered risk factors (meat origin, refined fats). Also, the oxidative-antioxidative balance will be evaluated by determining markers: oxidated glutathione/reducted glutathione, catalase enzyme, superoxide dismutase, glutathion peroxidase and malonyldialdehyde.

DETAILED DESCRIPTION:
A total of 300 patients with osteoarthritis will be included in the study. The objective of the study is to investigate the eating behaviour of the patients included in the study by using a semiquantitative questionnaire (frequency and quantity) by estimating the foods that are known to be protective for osteoarthritis (vegetables, fruits, cereals) as the ones that are considered risk factors (meat origin, refined fats). Also, the weight and height of each patient will be assessed and the patients will be included in 4 classes based on the body mass index: underweight, normal weight, overweight and obese. The type of physical activity will also be noted and the oxidative-antioxidative balance will be evaluated by determining serum markers: oxidated glutathione/reducted glutathione, catalase enzyme, superoxide dismutase, glutathion peroxidase and malonyldialdehyde. Correlation between eating behaviour, body mass index and oxidative stress markers will be made.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis
* signed informed consent

Exclusion Criteria:

* drugs or foods with antioxidant effects
* lack of judgement
* refuse to participate

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with osteoarthritis
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-07-17 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
serum concentration of oxidative stress markers | baseline
  oxidated glutathione/reduced glutathion, catalase enzyme, superoxide dismutase, glutathion peroxidase, malonyldialdehyde

CONTACTS AND LOCATIONS:
Overall Officials: Rodica A Ungur, MD, PhD, Principal Investigator — University of Medicine and Pharmacy Iuliu Hatieganu
Locations (1):
- Clinical Rehabilitation Hospital, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: Undecided
upon request